CLINICAL TRIAL: NCT05478941
Title: Can Virtual Reality Improve the Progressive Muscular Relaxation Technique Efficacy?
Acronym: VRelax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Caterina Novara, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4701
Record Dates: First submitted 2022-07-16; First posted 2022-07-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Coping Skills; Depression; Stress, Emotional; Quality of Life
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive Muscle Relaxation training via Zoom and Guided Imagery exposure (Active Comparator): A standardized protocol regarding the information on the training background is shared with participants. Then, they are invited to participate in four individual PMRT sessions (two sessions per week) deployed via Zoom.
  The fifth session after a week (T1; day 7) is administered in-presence at the Virtual Reality laboratory (A10-A11)- University of Padova; here an in-imagination relaxing scenario is built up with the support of the Psychotherapist; then, participants are exposed to an in-vivo PMRT relaxing session conducted by the Psychotherapist, with the request to think about the in-imagination relaxing scenario, created before, during the progressive relaxation procedure. After two weeks (T2; day 14), at the follow-up phase, the therapist asks to recover the in-imagination relaxing scenario and relax, giving participants the time allowed for the last guided relaxing session.
  Interventions: Behavioral: Progressive Muscular Relaxation via Zoom, and Exposure to a Guided Imagery Exposure.
- Progressive Muscle Relaxation training via Zoom and personalized VR exposure (Experimental): PMRT sessions and expected time length are the same as for the first group. Differences regard the fifth session after a week (T1; day 7), where the relaxing scenario is built with the psychotherapist's support based on the VR's tools. Indeed, during the in-presence session, participants are exposed to a merged personalized relaxing VR scenario and PMRT session administered by the Oculus Quest 2 tool.
  During the follow-up (T2; day 14), it is asked to recover the image and relax, making available the same time allowed for the last guided session.
  Interventions: Combination Product: Progressive Muscular Relaxation via Zoom, and Exposure to a Virtual Reality scenarios deployed by an Head mounted tool (Oculus Quest 2).
- Progressive Muscle Relaxation training based on audio-recording and personalized VR exposure (Experimental): A standardized protocol of information and the four PMRT sessions is administered individually based on an audio-track through the Moodle e-learning platform of the University of Padova.
  During the fifth session after a week (T1; day 7), users are asked to participate in an in-presence session in which they are exposed to a merged personalized, relaxing VR scenario and a PMRT session administered based on the Oculus Quest 2 tool. The last follow-up session (T2; day 14) has the same features as the other groups.
  Interventions: Combination Product: Progressive Muscular Relaxation via Audio-track, and Exposure to a Virtual Reality scenarios deployed by an Head mounted tool (Oculus Quest 2).

INTERVENTIONS:
Combination Product: Progressive Muscular Relaxation via Zoom, and Exposure to a Virtual Reality scenarios deployed by an Head mounted tool (Oculus Quest 2). — * Four individual PMRT sessions via Zoom.
  * In vivo PMRT relaxing session and Virtual Reality exposure (T1; day 7).
  * Follow-up phase (T2; day 14), after two weeks. Recovering the virtual reality scenario based on an in-imagination session, and the PMRT session.
  Arms: Progressive Muscle Relaxation training via Zoom and personalized VR exposure
Combination Product: Progressive Muscular Relaxation via Audio-track, and Exposure to a Virtual Reality scenarios deployed by an Head mounted tool (Oculus Quest 2). — * Four individual PMRT sessions via Audio-track.
  * In vivo PMRT relaxing session and Virtual Reality exposure (T1; day 7).
  * Follow-up phase (T2; day 14), after two weeks. Recovering the virtual reality scenario based on an in-imagination session, and the PMRT session.
  Arms: Progressive Muscle Relaxation training based on audio-recording and personalized VR exposure
Behavioral: Progressive Muscular Relaxation via Zoom, and Exposure to a Guided Imagery Exposure. — * Four individual PMRT sessions via Zoom.
  * In vivo PMRT relaxing session and Guided Imagery conducted by the Psychotherapist (T1; day 7).
  * Follow-up phase (T2; day 14), after two weeks. Recovering the in-imagination relaxing scenario and PMRT session.
  Arms: Progressive Muscle Relaxation training via Zoom and Guided Imagery exposure

SUMMARY:
The purposes of the current research project are as follows:

1. investigate if the PMRT associated with a personalized-relaxing scenario in VR can facilitate the recalling of the relaxing image in the real world than the standard procedure (consisting of PMRT associated with the in-imagination exposure to a comfortable subjective context). The investigators assume that VR would be more efficient than in-imagination since it would make easy the visualization process favor people cope with more realistic sensory experiences than in-imagination exposure. Accordingly, the VR exposure would elicit the strongest association between the relaxation procedure (neutral stimulus, NS) and the relaxing context in VR (conditioning stimulus, CS);
2. whether exposure to a personalized VREs has a more significant impact on anxiety, depression, stress, sense of presence, and quality of psychological well-being; these constructs are investigated by comparing the participants' performance on self-report questionnaires (described in the next section), before the start of the training (T0; baseline), at the end of all the four relaxing sessions, one week after the end of relaxation sessions (T1; day 7), and during follow up (T2; day 14);
3. if the relaxing sessions administered via Zoom are more proper for managing anxiety and stress than a procedure learned via an audio registration.

Considering the ability to generate vivid visual images is positively associated with the capacity to feel present in a virtual world, all the participants are asked to fulfill two questionnaires before the VR or the Guided Imagery exposure to investigate the vividness and the capacity to control mental images respectively, and to control the impact of these two dependent variables on the sense of presence self-reported after the in imagination or VR exposure.

DETAILED DESCRIPTION:
Each participant is randomly assigned to one of the three following different conditions:

1. Progressive Muscle Relaxation training via Zoom and Guided Imagery exposure A standardized protocol regarding the information on the training background is shared with participants.

   Then, they are invited to participate in four individually PMRT sessions (two sessions per week) deployed via Zoom.

   The fifth session (T1; day 7) is administered in-presence at the Virtual Reality Laboratory (A10-A11) - University of Padova; here, an in-imagination relaxing scenario is built up with the support of the Psychotherapist; then, participants are exposed to an in-vivo-PMRT-relaxing session conducted by the Psychotherapist, with the request to think about the in-imagination relaxing scenario, created before, during the progressive relaxation procedure.

   In the follow-up phase (T2, day 14), the therapist asks to recover the in-imagination relaxing scenario and relax, giving participants the same time allowed for the last guided relaxing session.
2. Progressive Muscle Relaxation training via Zoom and personalized VR exposure PMRT sessions and expected time length are the same as for the first group. Differences regard the fifth session, where the relaxing scenario is built with the psychotherapist support based on the VR's tools. Indeed, during the in-presence session, participants are exposed to a merged personalized and natural VR scenario and PMRT session administered by the Oculus Quest 2 tool.

   During the follow-up (T2; day 14), it is asked to recover the image and relax, making it available at the same time allowed for the last guided session.
3. Progressive Muscle Relaxation training based on audio-recording and personalized VR exposure In this condition, a standardized protocol of information and the four PMRT sessions are administered individually based on an audio track through the Moodle e-learning platform of the University of Padova.

During the fifth session (T1; day 7), users are asked to participate in an in-presence session in which they are exposed to a merged personalized, relaxing VR scenario and a PMRT session administered based on the Oculus Quest 2 tool. The last follow-up session has the same features as the other groups.

Assessment phases and Experimental procedure

T0 (baseline; before the PMRT sessions): 37 minutes.

The T0 assessment is the same for all participants and is administered at the Virtual Reality Laboratory (A10-A11)- Department of General Psychology, University of Padua. It implies the administration of the following measures:

* a demographic schedule (addressing age, gender, nationality, mother-tongue, marital status, years of school attendance, employment status, psychological problems/disorders, drugs use, medical conditions, neuromuscular issues, previous injures, previous experiences in relaxation practice or anxiety management training, or with Oculus);
* a series of self-report questionnaires investigating depression, anxiety, stress, quality of life, and distress coping strategies [State Trait Anxiety Inventory-Y (STAI-Y), Depression Anxiety Stress Scales-21 (DASS-21), Psychological General Well-Being Index (PGWBI), Coping Orientation to the Problems Experienced-Nuova Versione Italiana (COPE-NVI));
* resting heart rate detection with MiBand 2.

Before and after the four relaxing sessions administered remotely: 20 minutes globally.

Before and after each relaxation session, the personal level of tension is assessed using a 0 (no tension) to 10 (extreme tension level) scale; moreover, the state-anxiety level is evaluated based on the STAI-Y1.

The four-relaxation sessions are administered 2-3 days apart from each other for all three groups. The assessment phase is administered online based on the Moodle e-learning platform (University of Padova).

T1 phase (day 7): approximately 60 minutes. Before and after each relaxation session, subjects of tension and anxiety are assessed using a 0 (no tension) to 10 (extreme tension level) scale, and the state-anxiety level is evaluated based on the STAI-Y1.

Then, participants have been exposed to a PMRT session merged with a VR or a Guided Imagery procedure.

Before the in-imagination or the VR experience, all the participants fill out the Vividness of Visual Imagery Questionnaire (VVIQ) and the Test of Visual Imagery Control (TVIC). After the PMRT session, users compile a series of self-report questionnaires investigating depression, anxiety, stress, and quality of life (STAI-Y, DASS-21, PGWBI), and the VR group only fills out the VRSQ to monitor VR-related side effects (e.g., sickness, and headache), and the ITC-Sense of Presence Inventory to assess the sense of presence at the end of T1 phase.

The MiBand 2 was used during the entire T1 phase administration to detect the resting heart rate activity.

This assessment phase is administered based on the Moodle e-learning platform.

T2 (follow up; day 14): approximately 45 minutes. Before and after each relaxation session, subjects of tension and anxiety are assessed using a 0 (no tension) to 10 (extreme tension level) scale, and the state-anxiety level is evaluated based on the STAI-Y1.

All the users were exposed to a self-guided imagery experience in which those who were part of the VR group were asked to recall the personalized VR scenario experienced during the T1 phase (day 7). Instead, the Guided Imagery group retrieved the image participants had used in association with the PMRT during the T1 phase (day 7).

After the session, participants compile a series of self-report questionnaires investigating depression, anxiety, stress, quality of life (STAI-Y, DASS-21, PGWBI), and an ad hoc version based on the ITC-Sense of Presence Inventory to assess the sense of presence experienced during the imagery experience.

This assessment phase is administered based on the Moodle e-learning platform.

The follow-up assessment procedure requires approximately 25 minutes and is based on:

-a series of self-report questionnaires investigating depression, anxiety, stress, and quality of life (STAI-Y, DASS-21, PGWBI).

The MiBand 2 was used during the entire T1 phase administration (day 7), to detect the resting heart rate activity.

In general, the risks identified are principally related to difficulties in the technical implementation; in this context, mitigations strategies are represented by the feasibility study conducted in 2021, which helped obtain information for improving the VR environments according to users' needs and preferences. Effective recruitment strategies are deployed in the Trentino and Veneto regions to cope with the possible risk of drop-out of participants.

ELIGIBILITY:
Inclusion Criteria:

* General population
* Italian speaker
* Adult (age=> 18)
* Must be able to use a PC
* Must be able to use a Smartphone

Exclusion Criteria:

* Mental disorder diagnosis
* Clinical diagnosis of a neurological disorder
* Clinical diagnosis of epilepsy
* Have cardiac pacemakers
* Have metallic devices in the head-neck area
* Clinical diagnosis of infectious disorders
* Clinical diagnosis of gastrointestinal disorders
* Open wounds at the face level
* Clinical diagnosis of motor or visual dysfunctions
* Neuromuscular pain prevent the use of Oculus Quest 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with VR-related side effects as assessed by the Virtual Reality Sickness Questionnaire and the investigators' observations. | T1 (day 7)
  Participants in the two experimental arms is asked to refer if the VR head mounted display was painful, too heavy, or uncomfortable. More in detail, participants is asked if they have experienced negative side effect during the Virtual Reality (VR) exposure based on the Virtual Reality Sickness Questionnaire (VRSQ), administered at the end of the VR exposure. This questionnaire is based on a dichotomous answer (Yes/No). During the VR experience, the investigator observe participant reactions and record behaviors and signs suggesting an unpleasant experience.
Change is being assessed between and within subjects in depression scores | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in depression scores are assessed based on the "Depressive Anxiety Stress Scale-21-Depression subscale". Items are answered according on a 4-point Likert scale (0-3). Scores ranging from 0 to 42 (the scores will need to be multiplied by 2 to calculate the final score). Higher scores indicated more depression severity.
Change is being assessed between and within subjects in trait-anxiety scores | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in trait-anxiety scores are assessed based on the State-Trait Anxiety Inventory-Y2 (Trait Anxiety). The measure is a self-report questionnaire investigating the trait anxiety based on a 4-point Likert scale (1-4). Scores ranging from 20 to 80. Higher scores indicated higher trait-anxiety severity.
Change is being assessed between and within subjects in state-anxiety scores | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in state-anxiety scores are assessed based on the State-Trait Anxiety Inventory-Y1 (State anxiety) before and after each sessions. The STAI-Y1 is a self-report questionnaire investigating the state anxiety based on a 4-point Likert scale (1-4). Scores ranging from 20 to 80. Higher scores indicated more state-anxiety severity.
Change is being assessed between and within subjects in autonomic arousal, skeletal muscle effects, situational anxiety, subjective experience of anxious affect. | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in anxiety scores are assessed by the "Depressive Anxiety Stress Scale-21-Anxiety Subcale" based on a 4-point Likert scale (0-3). Scores ranging from 0 to 42 (the scores will need to be multiplied by 2 to calculate the final score). Higher scores indicated more anxiety severity.
Change is being assessed between and within subjects in bodily anxiety sensations | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in bodily anxiety sensations scores are assessed based on the Self Assessment Manikin (SAM). The SAM is a non-verbal imagery-based assessment technique used to assess bodily anxiety sensations that directly measures the pleasure, arousal, and dominance associated with a person's affective reaction to a wide variety of stimuli. Each sensations is assessed on 5 different images distributed in order of size. Participants can tick either of the five pictures or any of the four spaces in between, making it essentially a 9-point Likert-scale. The SAM varies from a minimum score of 3 to a maximum score of 27. The huge non-verbal imagery are related with higher bodily anxiety sensations.
Change is being assessed between and within subjects in levels of chronic non-specific arousal (stress) | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in levels of chronic nonspecific arousal (stress) scores are assessed by the "Depressive Anxiety Stress Scale-21-Stress subscale" based on a 4-point Likert scale (0-3). Scores ranging from 0 to 42 (the score will need to be multiplied by 2 to calculate the final score). Higher scores indicated higher level of stress.
Change is being assessed between and within subjects in relaxation levels | T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in relaxation levels are assessed based on the Visual Analog Scale administered before and after each sessions. This measure assess relaxation levels before and after each virtual reality experience. Participants had to express how relaxed they felt (0 =not at all relaxed; 10=completely relaxed; 0 =absent; 10=complete). Higher scores indicated higher relaxation levels.
Change is being assessed between and within subjects in quality of life scores | T0 (baseline), T1 (day 7), T2 (day 14)
  Change from baseline to T1 and T2 phases in quality of life scores on the Psychological General Well-Being Index are assessed at three different assessment times. The measure consists of 22 self-administered items, rated on a 6-point scale (0-5), which assess the psychological and general well-being. Scores ranging from 0 to 110. Higher scores indicated a better well-being state.
Change is being assessed between and within subjects in coping strategies scores | T0 (baseline), T1 (day 7), T2 (day 14)
  Change from baseline to T1 and T2 phases in coping strategies are assessed at three different assessment times. The Coping Orientation to the Problems Experienced-New Italian Version is a self-report questionnaire developed to assess the different coping strategies people use in response to stress; it is based on 60 items rated on a 4-point scale (1-4). Total scores ranging from 60 to 240. Higher scores indicate that a certain cope strategies is frequently used by the person.
Change is being assessed between and within subjects in sense of presence scores related to the Virtual Reality and Guided Imagery experiences | T1 (day 7), T2 (day 14)
  Differences between groups and change from T1 and T2 phases in sense of presence related to the VR or Guided Imagery experience are assessed at two different assessment times based on a Visual Analogue Scale and the ITC-Sense of Presence Inventory (ITC-SOPI). The ITC-SOPI is a self-report questionnaire assessing the sense of presence. Items are rated on a 5-point Likert scale (1-5). Scores ranging from 36 to 180. To obtain the scores for each of the scales, the average of the items have to be calculated. Higher scores indicated higher sense of presence.
Change is being assessed between and within subjects in hearth frequency | T0 (baseline), T1 (day 7), T2 (day 14)
  Differences between groups and change from baseline to T1 and T2 phases in hearth frequency are assessed based on the Xiaomi Mi Band 2 tool. It is used in three different assessment times (T0, T1, T2). During T1 and T2 hearth frequency is measured before, during, and after the in-presence relaxation session.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Novara, PhD, Principal Investigator — University of Padova
Locations (1):
- University of Padova, Padua, Italy

REFERENCES:
- [Derived] Pardini S, Gabrielli S, Olivetto S, Fusina F, Dianti M, Forti S, Lancini C, Novara C. Personalized Virtual Reality Compared With Guided Imagery for Enhancing the Impact of Progressive Muscle Relaxation Training: Pilot Randomized Controlled Trial. JMIR Ment Health. 2024 Jan 30;11:e48649. doi: 10.2196/48649. PMID 38289673
- [Derived] Pardini S, Gabrielli S, Olivetto S, Fusina F, Dianti M, Forti S, Lancini C, Novara C. Personalized, Naturalistic Virtual Reality Scenarios Coupled With Web-Based Progressive Muscle Relaxation Training for the General Population: Protocol for a Proof-of-Principle Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 17;12:e44183. doi: 10.2196/44183. PMID 37067881